CLINICAL TRIAL: NCT02517008
Title: Measuring the Impact of Non-monetary Incentives on Facility Delivery in Rural Zambia: A Clustered Randomized Controlled Trial
Brief Title: The Impact of Non-monetary Incentives on Facility Delivery in Rural Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDinsight (Other)
Collaborators: Ministry of Health, Zambia (Other Government); Minister of Community Development, Mother and Child Health, Zambia (Other); UNICEF (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 002
Record Dates: First submitted 2015-07-27; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Maternal Health
Keywords: non-monetary incentive; institutional delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mama kits intervention (Experimental): Health facilities randomized to this arm provided mama kits - packages of childcare materials including a cloth ("chitenge"), baby blanket, and diaper - to all mothers who delivered at these facilities between June 1, 2013 - Aug 31, 2013.
  Interventions: Other: Mama kit
- No intervention (No Intervention): Health facilities randomized to this arm provided obstetric services as normal.

INTERVENTIONS:
Other: Mama kit — A low-cost non-monetary incentive (mama kit) was provided to all women who delivered at the facility between June 1, 2013 - Aug 31, 2013. Women were told about the intervention during ANC, and safe motherhood groups in the community promoted the intervention in the catchment areas of the treatment facilities.
  Arms: Mama kits intervention

SUMMARY:
This study measured the impact and cost-effectiveness of a low-cost, non-monetary incentive ("mama kit") on rural facility delivery rates in Zambia.

DETAILED DESCRIPTION:
This clustered randomized controlled trial assessed the impact of providing a package of childcare items (a cloth, baby diaper, and blanket) to women conditional upon delivering at a facility on facility delivery rates in rural Serenje and Chadiza Districts in Zambia. Facilities were randomized to either provide the intervention or not. Facility-level antenatal care (ANC) and delivery registers were used to measure the percentage of women attending antenatal care who delivered at a study facility during the intervention period. Results from the trial were then used to model the cost-effectiveness of mama kits at-scale in terms of cost per death averted.

ELIGIBILITY:
Inclusion Criteria:

* Had an antenatal care record at one of the study facilities
* Had an estimated date of delivery (as measured by estimated date of last menstrual period, estimated date of delivery, or estimated gestational age in weeks as recorded in the antenatal care register) between June 1, 2013 - Aug 31, 2013.

Exclusion Criteria:

* Did not have an antenatal care record at one of the study facilities
* Had an estimated date of delivery outside of the intervention window (June 1, 2013 - Aug 31, 2013)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2159 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Facility delivery ratios | At delivery, up to 10 months after the first antenatal care visit date
  Administrative data were used to measure the outcome. Antenatal care and delivery records were linked across registers. Women who had attended ANC and were linked to a record in the registry was counted as having delivered at a facility.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, MPAID/MBA, Principal Investigator — IDinsight